CLINICAL TRIAL: NCT03120429
Title: Effects of Moderate Consumption Lean Fish on Weight Loss of Overweight and Obese Women During a Weight Loss Program, a 24 Week Randomized Controlled Trial
Brief Title: Effects of Moderate Consumption of Lean Fish on Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novindiet Clinic (Other)
Collaborators: University of Nottingham (Other); Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ND-203
Record Dates: First submitted 2017-04-15; First posted 2017-04-19 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Obesity; Overweight
Keywords: lean fish; weight loss; Diet
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fish group (Experimental): subjects will have 3 x 150 g lean fish/ week at main meal
  Interventions: Behavioral: Fish group
- Control group (Experimental): subjects will have no seafood.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Fish group — Fish group will have hypoenergetic diet in which subjects will have 3 x 150 g lean fish/ week at main meal
  Other Names: FG
  Arms: Fish group
Behavioral: Control group — Control group will have hypo-energetic diet in which subjects have no seafood.
  Other Names: CG
  Arms: Control group

SUMMARY:
the aim of present study is to compare the specific effects moderate consumption of lean fish on weight loss of healthy obese and overweight female adults, while participants follow energy-restricted diets also to investigate the effects of this intervention on carbohydrate and lipid profiles, as cardiometabolic risk factors.

ELIGIBILITY:
Inclusion Criteria:

* female
* 18-45 years of age.
* Body mass index (BMI) between 27.5-35 kg/m²
* Must be able to have moderate exercise.
* Must be interested to lose weight

Exclusion Criteria:

* Pregnancy or lactation during the previous 6 months, or planned pregnancy in the next six months.
* Taking medications that could affect metabolism or change body weight.
* Report heart problems, chest pain, and cancer within the last five years.
* Use of supplements containing n-3 fatty acids, calcium or vitamin-D during the last 3 months.
* Consumption of fish and sea foods regularly
* Smoking
* Menopause
* Diagnosis of any chronic disease such as fatty liver, cancer, chemo/radio therapy, heart disease, immune compromised conditions, abnormal thyroid hormone level.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-25 (Actual); Primary Completion 2019-01-22 (Actual); Study Completion 2019-10-13 (Actual)

PRIMARY OUTCOMES:
weight loss | 24 Weeks
  kg

SECONDARY OUTCOMES:
waist circumference | 24 Weeks
  cm
fasting plasma glucose | 24 Weeks
  mmol/l
serum insulin level | 24 Weeks
  mU/l
insulin resistance (HOMA-IR) | 24 Weeks
  score
glycosylated hemoglobin (HbA1c) | 24 Weeks
  percentage (%)
lipid profiles | 24 Weeks
  mmol/l
liver enzymes (SGOT, SGPT) | 24 Weeks
  U/l

CONTACTS AND LOCATIONS:
Locations (1):
- NovinDiet Clinic, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided